CLINICAL TRIAL: NCT01610440
Title: Phase I/II Study of Stem Cell Therapy in Patients With Duchenne Muscular Dystrophy
Brief Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Therapy for Patients With Duchenne Muscular Dystrophy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Beike Bio-Technology Co., Ltd. (Industry)
Collaborators: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BKCR-DMD-1(Ⅰ)
Record Dates: First submitted 2012-05-21; First posted 2012-06-04 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Human Umbilical Cord Mesenchymal Stem Cells
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Group (Experimental): Participants will be given rehabilitation therapy plus human umbilical cord mesenchymal stem cells transplantation with one year follow-up
  Interventions: Biological: human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cells — rehabilitation therapy plus human umbilical cord mesenchymal stem cells

SUMMARY:
Duchenne muscular dystrophy (DMD), an X-linked recessive genetic disease always progressed slowly，tends to leading proximal skeletal muscle atrophy and weakness of limbs, as well as impaired respiratory muscle and cardiac muscle. To a large extent, patients always lose motor function gradually and die for heart failure or severe infection at the end stage of DMD. At present, the treatment strategy relies on heteropathy accompanied with rehabilitation training. However, the therapeutic effect remains extremely limited.

Human umbilical cord mesenchymal stem cells (hUC-MSCs) have been evidenced to improve motor function, increase muscle strength and reduce abnormal levels of related enzymes, such as creatine kinase (CK), lactate dehydrogenase (LDH), alanine aminotransferase (ALT) and aspartate aminotransferase (AST). This study is aimed to explore the safety and efficacy of hUC-MSCs transplantation for DMD.

DETAILED DESCRIPTION:
This study is designed to investigate the safety and efficacy of human umbilical cord mesenchymal stem cells transplantation in patients with progressive muscular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5-12 years
* Clinical manifestation, enzymology, electromyogram, gene type confirmed the diagnose of Duchenne muscular dystrophy
* Sign the consent form and follow the clinic trail procedure

Exclusion Criteria:

* Not Duchenne muscular dystrophy
* Any history of hypersensitivity to serum products,or other know drug and food allergy
* Combined Pneumonia or other Severe systemic bacteria infection
* HIV+, TPPA +， patients diagnosed as HBV or HCV
* Tumor Markers +
* Severe psychotic patients, cognitive dysfunction
* Coagulation disorders
* Uncontrolled hypertension after treatment，blood pressure≥180mmHg/110 mmHg
* Other severe systemic or organic disease
* Enrollment in other trials in the last 3 months
* Received any stem cell therapy in past 6 months
* Other criteria that investigator consider improper for inclusion

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-03 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Activities of Daily Living(ADL)scale | 1 year after treatment

SECONDARY OUTCOMES:
Incidences of Adverse Event and Serious Adverse Event | 1 year after treatment
Change from baseline in CK | 1 year after treatment
Change from baseline in LDH | 1 year after treatment
Change from baseline in ALT | 1 year after treatment
Change from baseline in AST | 1 year after treatment
Change from baseline to manual muscle test(MMT) | 1 year after treatment
Change from baseline in electromyography(EMG) | 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Liqing Yao, Principal Investigator — The Second Affiliated Hospital of Kunming Medical University
Locations (1):
- The Second Affiliated Hospital of Kunming Medical College, Kunming, Yunnan, China